CLINICAL TRIAL: NCT06231550
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Axl Inhibitor FC084CSA in Patients With Advanced Malignant Solid Tumors
Brief Title: A Study of Axl Inhibitor FC084CSA in Patients With Advanced Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FindCure Biosciences (ZhongShan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FC084-CA-101
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Advanced Malignant Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FC084CSA (Experimental)
  Interventions: Drug: FC084CSA tablets

INTERVENTIONS:
Drug: FC084CSA tablets — FC084CSA accelerated doses at 100mg QD, and then started the conventional "3+3" design from 200mg QD.

SUMMARY:
This is a phase I clinical study to evaluate safety, tolerability, pharmacokinetic characteristics and preliminary efficacy of Axl inhibitor FC084CSA in patients with advanced malignant solid tumors who have failed standard anti-cancer treatment.

DETAILED DESCRIPTION:
FC084CSA accelerated doses at 100mg QD, and then started the conventional "3+3" design from 200mg QD.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years old male and female.
2. Patients with advanced malignant solid tumors who have failed standard treatments.
3. According to RECIST 1.1, there is at least one measurable lesion.
4. ECOG performance status 0-1.
5. Laboratory examination should meet: ① Blood routine: hemoglobin (HGB) ≥85 g/L, neutrophil count (ANC) ≥1.5×10^9/L, platelet count ( PLT) ≥75×10^9/L; ②Blood biochemistry: total bilirubin (TBIL) ≤1.5×upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0×ULN, serum creatinine ( Cr)≤1.5×ULN or calculate the creatinine clearance ≥50 mL/min according to the Cockcroft-Gault formula method.

Exclusion Criteria:

1. Not recovered from the adverse reactions caused by previous anti-tumor treatments (≥CTCAE grade 1).
2. Received anti-tumor therapy within 4 weeks before enrollment.
3. Participated in other clinical trials within 4 weeks before enrollment and used clinical investigational drugs during this period.
4. Have undergone surgery within 4 weeks before enrollment, and the investigator believes that the patient's state has not recovered to the point where the study can be started.
5. Patients with ascites (ascites), pleural effusion (pleural effusion) or pericardial effusion that cannot be controlled by drainage or other methods.
6. Central nervous system metastases with clinical symptoms.
7. With any situations that the researcher considers inappropriate to participate in this research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Determine the Maximum Tolerated Dose (MTD) | Approximately 12 months
  The highest dose is defined at which no more than 1 of 3 evaluable participants has had a Dose Limiting Toxicity (DLT) according to NCI CTCAE V5.0 criteria and determination by Investigator and Data and Safety Monitoring Committee.
Determine the Recommended Phase 2 Dose (RP2D) | Approximately 12 months
  The RP2D is based upon the review of all available data including safety, pharmacokinetic, preliminary anti-tumor activity, and MTD.
Determine dose-limiting toxicity (DLT) | 24 days after first dose
  Determine the DLT of FC084CSA
Frequency of adverse events (AEs) and SAEs | Approximately 12 months
  To investigate the safety characteristics of FC084CSA

SECONDARY OUTCOMES:
Objective response rate (ORR) | Approximately 12 months
  To explore the clinical effectiveness. Tumor response based on RECIST 1.1
Disease control rate (DCR) | Approximately 12 months
  DCR as assessed using RECIST 1.1
Progression free survival (PFS) | Approximately 12 months
  PFS as assessed using RECIST 1.1
Pharmacokinetic (PK) Cmax | Approximately 12 months
  To investigate the pharmacokinetic (PK) profile of FC084CSA
Pharmacokinetic (PK) Tmax | Approximately 12 months
  To investigate the pharmacokinetic (PK) profile of FC084CSA
Pharmacokinetic (PK) AUC 0-t | Approximately 12 months
  To investigate the pharmacokinetic (PK) profile of FC084CSA
Pharmacokinetic (PK) AUC 0-∞ | Approximately 12 months
  To investigate the pharmacokinetic (PK) profile of FC084CSA
Pharmacokinetic (PK) t1/2 | Approximately 12 months
  To investigate the pharmacokinetic (PK) profile of FC084CSA

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No